CLINICAL TRIAL: NCT07327710
Title: Efficacy and Safety of Non-Invasive Brain-Computer Interface Combined With Transcranial Electrical Stimulation in the Treatment of Peripheral Facial Palsy
Brief Title: Non-Invasive Brain-Computer Interface Combined With Transcranial Electrical Stimulation for Peripheral Facial PalsyStimulation in the Treatment of Peripheral Facial Palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fang Liu, phD, Nanjing Medical University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: [2025]YLJSA075
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Facial Palsy; Pulsed Radiofrequency; Brain-Computer Interface; Transcranial Direct Current Stimulation
MeSH Terms: interventions — Brain-Computer Interfaces; Transcranial Direct Current Stimulation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Standard Therapy (Placebo Comparator): Standard therapy.
  Interventions: Other: Standard Therapy
- Group B: Pulsed Radiofrequency + Standard Therapy (Placebo Comparator): Standard Therapy and Pulsed Radiofrequency Therapy.
  Interventions: Procedure: Pulsed Radiofrequency （PRF）; Other: Standard Therapy
- Group C：BCI + tDCS + Pulsed Radiofrequency Treatment + Standard Therapy (Experimental): BCI + tDCS + Pulsed Radiofrequency Treatment + Standard Therapy.
  Interventions: Procedure: Brain-Computer Interface （BCI）; Procedure: Pulsed Radiofrequency （PRF）; Other: Standard Therapy

INTERVENTIONS:
Procedure: Brain-Computer Interface （BCI） — 1. BCI Therapy:
     Real-time feedback drives NMES (neuromuscular electrical stimulation) of the target facial muscles.
     Each session lasts 30 minutes, 3-5 times per week, for a total of 4 weeks.
  2. tDCS Therapy: Applied to the regions corresponding to the branches of the facial nerve. A constant current (usually 0.5-2 mA) is delivered for 20-30 minutes per session, 5-20 sessions per course.
  Standard treatment frequency is once daily, 5-6 times per week, with a continuous course of 2-4 weeks. Each stimulation session typically lasts 20-30 minutes.
  Other Names: transcranial Direct Current Stimulation （tDCS）
  Arms: Group C：BCI + tDCS + Pulsed Radiofrequency Treatment + Standard Therapy
Procedure: Pulsed Radiofrequency （PRF） — Acute-phase "shock" protocol: Within 7 days of onset, a single pulsed radiofrequency treatment is applied to the extracranial segment of the facial nerve. Depending on recovery, the treatment may be repeated 1-2 weeks later.
  Chronic-phase (sequelae) "shock" protocol: Administered once every 1-4 weeks, for a total of 1-4 sessions.
  Arms: Group B: Pulsed Radiofrequency + Standard Therapy; Group C：BCI + tDCS + Pulsed Radiofrequency Treatment + Standard Therapy
Other: Standard Therapy — Includes facial muscle function training, physiotherapy, hot and cold compresses, and neurotrophic drug treatment.

SUMMARY:
To evaluate the efficacy and safety of treating peripheral facial palsy using a non-invasive brain-computer interface combined with transcranial direct current stimulation (tDCS).

DETAILED DESCRIPTION:
This study is mainly designed to compare the therapeutic efficacy of non-invasive brain-computer interface combined with transcranial direct current stimulation (tDCS), pulsed radiofrequency, and pharmacological treatment versus pulsed radiofrequency combined with pharmacological treatment in patients with peripheral facial palsy.

ELIGIBILITY:
Inclusion Criteria:

Aged 18-70 years, regardless of sex.

Unilateral peripheral facial nerve palsy.

House-Brackmann (HB) grade II-VI.

Able to cooperate with target facial movement tasks and provide written informed consent, with intact cognitive function and good communication ability.

Good skin condition, with no severe skin lesions or facial skin grafts; no implanted electronic devices such as cardiac pacemakers or deep brain stimulators, to avoid electrophysiological interference.

Non-pregnant and non-lactating women, in accordance with regulatory requirements for minimal-risk research.

Exclusion Criteria:

Open facial wounds, active infections, significant skin lesions, or a history of severe allergy.

Severe cognitive impairment, psychiatric disorders, or inability to comply with study procedures.

Occurrence of serious adverse events or withdrawal at the patient's request.

Pregnant or lactating women, or patients unable to use appropriate contraceptive measures during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in House-Brackmann (HB) grading | At 0，2，4，8 and 12 weeks.
Sunnybrook Facial Grading System score. | At 0，2，4，8 and 12 weeks.
Static and dynamic facial symmetry scores. | At 0，2，4，8 and 12 weeks.
Degree of facial muscle EMG activation and changes in EEG functional connectivity. | At 0，2，4，8 and 12 weeks.

SECONDARY OUTCOMES:
Adverse events | At 0，2，4，8 and 12 weeks.
  Adverse events included skin tingling at the electrode site, mild fatigue, burning sensation, itching, headache, and a potential risk of seizure induction.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Peoples's Hospital of Changzhou, the Third Affiliated Hospital of Nanjing Medical University, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because the study involves sensitive clinical and neurophysiological data, and full de-identification cannot be guaranteed without compromising participant privacy. In addition, the informed consent obtained from participants did not include provisions for public data sharing.

REFERENCES:
- [Result] Soekadar SR, Witkowski M, Birbaumer N, Cohen LG. Enhancing Hebbian Learning to Control Brain Oscillatory Activity. Cereb Cortex. 2015 Sep;25(9):2409-15. doi: 10.1093/cercor/bhu043. Epub 2014 Mar 13. PMID 24626608
- [Result] Jitsinthunun T, Li C, Ng TK, Zinboonyahgoon N. Pulsed Radiofrequency Treatment: Evidence for and Applications in Chronic Pain. Pain Physician. 2025 Nov;28(6):467-481. PMID 41337760
- [Result] Sam J, Catapano M, Sahni S, Ma F, Abd-Elsayed A, Visnjevac O. Pulsed Radiofrequency in Interventional Pain Management: Cellular and Molecular Mechanisms of Action - An Update and Review. Pain Physician. 2021 Dec;24(8):525-532. PMID 34793641
- [Result] Liu Z, Xie D, Wen X, Wang R, Yang Q, Liu H, Shao Y, Liu T. Peripheral Repetitive Transcranial Magnetic Stimulation(rTMS) for Idiopathic Facial Nerve Palsy: A Prospective, Randomized Controlled Trial. Neural Plast. 2022 Jul 13;2022:7536783. doi: 10.1155/2022/7536783. eCollection 2022. PMID 35875789
- [Result] Li D, Li R, Song Y, Qin W, Sun G, Liu Y, Bao Y, Liu L, Jin L. Effects of brain-computer interface based training on post-stroke upper-limb rehabilitation: a meta-analysis. J Neuroeng Rehabil. 2025 Mar 3;22(1):44. doi: 10.1186/s12984-025-01588-x. PMID 40033447
- [Result] Cervera MA, Soekadar SR, Ushiba J, Millan JDR, Liu M, Birbaumer N, Garipelli G. Brain-computer interfaces for post-stroke motor rehabilitation: a meta-analysis. Ann Clin Transl Neurol. 2018 Mar 25;5(5):651-663. doi: 10.1002/acn3.544. eCollection 2018 May. PMID 29761128
- [Result] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Corrigendum to "Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018)" [Clin. Neurophysiol. 131 (2020) 474-528]. Clin Neurophysiol. 2020 May;131(5):1168-1169. doi: 10.1016/j.clinph.2020.02.003. Epub 2020 Feb 19. No abstract available. PMID 32122766